CLINICAL TRIAL: NCT02242201
Title: Prospective, Randomized Controlled Trial Comparing Continuous Posterior Lumbar Plexus Nerve Block vs Periarticular Injection With Ropivacaine or Liposomal Bupivacaine (Exparel®) on Patients Undergoing Total Hip Arthroplasty
Brief Title: Total Hip Arthroplasty (THA) Lumbar Plexus Verses Periarticular
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rebecca L Johnson, MD, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-004183; UL1TR000135 (NIH)
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Bupivacaine; Ropivacaine; Epinephrine; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PNB Bupivacaine (Active Comparator): Bupivacaine 0.5% with 1:200,000 epinephrine 30 ml bolus preoperatively followed by an infusion of bupivacaine 0.2% on post anesthesia care unit (PACU) arrival.
  Interventions: Drug: PNB Bupivacaine; Drug: Epinephrine
- PAI Ropivacaine (Active Comparator): Patients 50 to 74.9 kg: ropivacaine 200 mg, epinephrine 100 ug, ketorolac 30 mg. Patients 75 to 99.9 kg: ropivacaine 300 mg, epinephrine 200 ug, ketorolac 30 mg. Patients 100 to 125 kg: ropivacaine 400 mg, epinephrine 300 ug, ketorolac 30mg.
  Interventions: Drug: PAI Ropivacaine; Drug: Epinephrine; Drug: Ketorolac
- PAI liposomal bupivacaine (Active Comparator): Liposomal bupivacaine 255 mg, ketorolac 30 mg, bupivacaine 125 mg, epinephrine 125 ug.
  Interventions: Drug: PAI liposomal bupivacaine; Drug: Epinephrine; Drug: Ketorolac

INTERVENTIONS:
Drug: PNB Bupivacaine — Infusion
  Other Names: Marcaine
  Arms: PNB Bupivacaine
Drug: PAI Ropivacaine — Injection
  Other Names: Naropin
  Arms: PAI Ropivacaine
Drug: PAI liposomal bupivacaine — Injection
  Other Names: Exparel
  Arms: PAI liposomal bupivacaine
Drug: Epinephrine — Injection, weight-based dosage of 100 mcg - 300 mcg
Drug: Ketorolac — Injection, 30 mg
  Other Names: Acuvail; Acular
  Arms: PAI Ropivacaine; PAI liposomal bupivacaine

SUMMARY:
Total hip arthroplasty is a one of the most commonly performed surgical procedures with increasing numbers anticipated over the next several decades. The purpose of this study was to find a better way to make patients comfortable after their hip surgery. Three different ways of providing pain relief were compared, a peripheral nerve block in the lower back outside of the spinal space (using bupivacaine, a numbing medicine), or injections around the hip joint with one of two different medicines, either Ropivacaine or Liposomal Bupivacaine (Exparel®).

DETAILED DESCRIPTION:
Total hip arthroplasty is associated with moderate to severe postoperative pain and an ideal clinical pathway for pain management has yet to be established. Multimodal pain management incorporating the use of regional anesthesia for THA has led to decreased hospital length of stay, improved patient comfort, and enhanced patient satisfaction that is efficacious and cost-effective. This investigation compared multimodal total joint arthroplasty pathways with continuous lumbar plexus blockade versus two different periarticular injection mixtures to potentially determine an ideal perioperative analgesia pathway for THA.

Patients undergoing elective, unilateral primary total hip arthroplasty within a clinical pathway utilizing preemptive low-dose opioid and non-opioid medications for multimodal analgesia were randomized to one of three different intervention groups after informed consent was obtained: posterior lumbar plexus block (PNB), periarticular infiltration (PAI) with ropivacaine, ketorolac, and epinephrine, and PAI with liposomal bupivacaine, ketorolac, and epinephrine. The investigators hypothesized differences in the analgesia outcomes between the three intervention groups would provide for an evidenced-based clinical pathway to emerge as a result of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III
2. Patients presenting for unilateral primary total hip arthroplasty
3. Patients 18 years of age and older

Exclusion Criteria:

1. Chronic pain syndromes such as fibromyalgia or complex regional pain syndrome
2. History of long term use of daily opioids (>1 months) with Oral Morphine Equivalent (OME) >5mg/day
3. Body mass index (BMI) > 40 kg/m2
4. Allergies to medications used in this study such as: fentanyl,hydromorphone, ketorolac, ibuprofen, acetaminophen, local anesthetics, oxycodone, tramadol, ondansetron, droperidol, dexamethasone, celecoxib and OxyContin
5. Major systemic medical problems such as:

   1. severe renal disorder defined as glomerular filtration rate (GFR) <50 units/m2
   2. cardiovascular disorders defined as Congestive Heart Failure (CHF) New York Heart Association (NYHA) class III-IV
   3. severe hepatic disorder defined as current or past diagnosis of acute/subacute necrosis of liver, acute hepatic failure, chronic liver disease, cirrhosis (primary biliary cirrhosis), fatty liver, chronic hepatitis/toxic hepatitis, liver abscess, hepatic coma, hepatorenal syndrome, other disorders of liver
6. Impaired cognitive function or inability to understand the study protocol
7. Contraindication to a regional anesthesia technique (e.g., preexisting neuropathy in the operative extremity, coagulopathy [platelets < 100,000, International Normalized Ratio (INR) >1.5], refusal, etc.).
8. Previous contralateral hip replacement managed with regional or periarticular injection
9. Unable to follow-up at the 3 month interval at Mayo Clinic in Rochester, Minnesota
10. Pregnancy or breastfeeding (women of child-bearing potential will require a negative pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Johnson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Johnson RL, Amundson AW, Abdel MP, Sviggum HP, Mabry TM, Mantilla CB, Schroeder DR, Pagnano MW, Kopp SL. Continuous Posterior Lumbar Plexus Nerve Block Versus Periarticular Injection with Ropivacaine or Liposomal Bupivacaine for Total Hip Arthroplasty: A Three-Arm Randomized Clinical Trial. J Bone Joint Surg Am. 2017 Nov 1;99(21):1836-1845. doi: 10.2106/JBJS.16.01305. PMID 29088038

RESULTS

PARTICIPANT FLOW:
Groups:
- PNB Bupivacaine: Bupivacaine 0.5% with 1:200,000 epinephrine 30 ml bolus preoperatively followed by an infusion of bupivacaine 0.2% on post anesthesia care unit (PACU) arrival.
  Posterior lumbar plexus block (PNB) Bupivacaine: Infusion
  Epinephrine: Injection, weight-based dosage of 100 mcg - 300 mcg
- PAI Ropivacaine: Patients 50 to 74.9 kg: ropivacaine 200 mg, epinephrine 100 ug, ketorolac 30 mg. Patients 75 to 99.9 kg: ropivacaine 300 mg, epinephrine 200 ug, ketorolac 30 mg. Patients 100 to 125 kg: ropivacaine 400 mg, epinephrine 300 ug, ketorolac 30mg.
  Periarticular infiltration (PAI) Ropivacaine: Injection
  Epinephrine: Injection, weight-based dosage of 100 mcg - 300 mcg
  Ketorolac: Injection, 30 mg
Period: Overall Study
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Started | 55 | 55 | 55
Completed | 51 | 54 | 54
Not Completed | 4 | 1 | 1
Not completed — preoperative identified neuropathy | 2 | 0 | 0
Not completed — planned post-op anticoagulation | 1 | 0 | 0
Not completed — changed surgical procedure | 1 | 0 | 0
Not completed — postponed surgery | 0 | 0 | 1
Not completed — preoperative opioid consumption | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine | Total
Number analyzed (Participants) | 51 | 54 | 54 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.5) | 59.4 (15.3) | 61.7 (11.7) | 61.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 28 | 80
  Male | 26 | 27 | 26 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 54 | 54 | 159
Duration of surgery [Mean (Standard Deviation); unit: minutes] | 91.4 (24.0) | 88.1 (23.2) | 88.4 (28.3) | 89.2 (25.2)
Type of anesthetic [Count of Participants; unit: Participants]
  General | 13 | 10 | 13 | 36
  Spinal | 38 | 44 | 41 | 123
American Society of Anesthesiologists (ASA) Status [Count of Participants; unit: Participants] — The ASA Physical Status Classification System assesses the fitness of patients prior to surgery. It defines an ASA I as a normal healthy patient, ASA II as a patient with mild systemic disease, and ASA III as a patient with severe systemic disease.
  Participants
    I or II | 44 | 41 | 45 | 130
    III | 7 | 13 | 9 | 29
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.0 (6.0) | 30.1 (6.0) | 30.2 (5.4) | 30.1 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Postoperative Pain Score
Description: Pain was measured on an ascending numeric rating scale (NRS) from 0-10 where 1-3 equaled mild pain, 4-6 equaled moderate pain, 7-9 equaled severe pain, and 10 equaled worst possible pain.
Time Frame: Post-Operative Day 1 (0600-1200)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 51 | 54 | 54
units on a scale | 3.0 [1 to 4] | 4.0 [2 to 5] | 3.0 [2 to 5]
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine; Test type: Superiority; p = 0.033, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; Test type: Superiority; p = 0.662, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; Test type: Superiority; p = 0.103, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Opioid Consumption During Hospitalization
Description: Measured in daily oral morphine equivalents (OME)
Time Frame: Preoperative, Intraoperative, Postanesthesia Care Unit (PACU), Post Operative Day (POD) 0, day 1, and day 2
Population: For Post Operative Day (POD) 2, data were missing for 26 subjects (7 in the PNB group, 9 in the PAI-R group, and 10 in the PAI-L group).
Measure: Median (Inter-Quartile Range); unit: Oral morphine equivalent in milligrams
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 51 | 54 | 54
Oral morphine equivalent in milligrams
  Preoperative | 15 [0 to 30] | 15 [0 to 30] | 15 [15 to 30]
  Intraoperative | 10 [5 to 20] | 10 [5 to 15] | 10 [5 to 20]
  Postanesthesia Care Unit (PACU) | 0 [0 to 10] | 0 [0 to 0] | 0 [0 to 10]
  Post Operative Day (POD) 0 post PACU | 7.5 [0 to 30] | 15 [0 to 30] | 11.3 [0 to 22.5]
  POD 1 | 22.5 [7.5 to 60] | 33.8 [7.5 to 60] | 15 [7.5 to 45]
  POD 2: number analyzed (Participants) | 44 | 45 | 44
  POD 2 | 15 [0 to 30] | 15 [0 to 45] | 11.3 [0 to 18.8]
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine; Preoperative; Test type: Superiority; p = 0.948, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; Preoperative; Test type: Superiority; p = 0.880, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; Preoperative; Test type: Superiority; p = 0.802, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: PNB Bupivacaine vs PAI Ropivacaine; Intraoperative; Test type: Superiority; p = 0.179, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; Intraoperative; Test type: Superiority; p = 0.837, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; Intraoperative; Test type: Superiority; p = 0.142, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: PNB Bupivacaine vs PAI Ropivacaine; PACU; Test type: Superiority; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; PACU; Test type: Superiority; p = 0.516, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; PACU; Test type: Superiority; p = 0.052, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: PNB Bupivacaine vs PAI Ropivacaine; POD 0 post PACU; Test type: Superiority; p = 0.840, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; POD 0 post PACU; Test type: Superiority; p = 0.744, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; POD 0 post PACU; Test type: Superiority; p = 0.501, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: PNB Bupivacaine vs PAI Ropivacaine; POD 1; Test type: Superiority; p = 0.358, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; POD 1; Test type: Superiority; p = 0.536, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; POD 1; Test type: Superiority; p = 0.110, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: PNB Bupivacaine vs PAI Ropivacaine; POD 2; Test type: Superiority; p = 0.313, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: PNB Bupivacaine vs PAI Liposomal Bupivacaine; POD 2; Test type: Superiority; p = 0.893, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: PAI Ropivacaine vs PAI Liposomal Bupivacaine; POD 2; Test type: Superiority; p = 0.232, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Hospital Length of Stay
Description: Discharge readiness was evaluated by the surgical team during morning and afternoon physical therapy sessions.
Time Frame: Post-operative Day 1 through discharge (approximately 3 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 51 | 54 | 54
days | 2 [2 to 2] | 2 [2 to 3] | 2 [2 to 2]
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Test type: Superiority; p = 0.772, Kruskal-Wallis

4. Other Pre Specified Outcome: Change in Unipedal Stance Time
Description: Length of time in seconds a patient could stand on involved leg
Time Frame: Baseline, 3 months
Population: Data were available for 50, 54, and 51 patients in the PNB, PAI Ropivacaine, and PAI liposomal bupivacaine groups, respectively.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 54 | 51
seconds
  Baseline | 24.5 [6 to 30] | 30 [9 to 30] | 30 [7 to 30]
  3 months | 30 [12 to 30] | 30 [18 to 30] | 30 [15 to 30]
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Baseline; Test type: Superiority; p = 0.251, Regression, Cox
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; 3 month follow-up; Test type: Superiority; p = 0.300, Regression, Cox
Statistical Analysis 3: Comparison: PNB Bupivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.113, Regression, Cox
Statistical Analysis 4: Comparison: PAI Ropivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.147, Regression, Cox
Statistical Analysis 5: Comparison: PAI Liposomal Bupivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.216, Regression, Cox
Statistical Analysis 6: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.968, Regression, Cox

5. Other Pre Specified Outcome: Post-Operative Pain Score
Description: Pain intensity (NRS) assessment at 3 month follow-up. Pain was measured on an ascending numeric rating scale (NRS) from 0-10 where 1-3 equaled mild pain, 4-6 equaled moderate pain, 7-9 equaled severe pain, and 10 equaled worst possible pain.
Time Frame: 3 month follow-up
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 54 | 51
units on a scale
  Pain at rest | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Pain with movement | 0 [0 to 1] | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Pain at rest; Test type: Superiority; p = 0.776, Kruskal-Wallis
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Pain with movement; Test type: Superiority; p = 0.447, Kruskal-Wallis

6. Other Pre Specified Outcome: Change in Short Form-36 (SF-36) Quality of Life Physical Component
Description: Scores on the Medical Outcomes Study 36-Item Short-Form General Health Survey (SF-36). Subjects completed the SF-36 which consists of 8 sub-scales ranging from 0 to 100, with (0 = worst imaginable, 100 = best imaginable).
Time Frame: Baseline, 3 months
Population: Data were available for 50, 52, and 51 patients in the PNB, PAI Ropivacaine, and PAI liposomal bupivacaine groups, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 52 | 51
units on a scale | 12.5 (10.3) | 12.6 (9.1) | 12.3 (8.8)
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Test type: Superiority; p = 0.986, ANOVA
Statistical Analysis 2: Comparison: PNB Bupivacaine; Baseline vs 3 months; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: PAI Ropivacaine; Baseline vs 3 months; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: PAI Liposomal Bupivacaine; Baseline vs 3 months; Test type: Superiority; p < 0.001, t-test, 1 sided

7. Other Pre Specified Outcome: Change in Short Form-36 (SF-36) Quality of Life Mental Component
Description: as for outcome 6
Time Frame: Baseline, 3 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 52 | 51
units on a scale | 2.2 (9.5) | 2.6 (9.4) | 3.0 (9.4)
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Test type: Superiority; p = 0.898, ANOVA
Statistical Analysis 2: Comparison: PNB Bupivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.112, t-test, 1 sided
Statistical Analysis 3: Comparison: PAI Ropivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.046, t-test, 1 sided
Statistical Analysis 4: Comparison: PAI Liposomal Bupivacaine; Baseline vs 3 months; Test type: Superiority; p = 0.026, t-test, 1 sided

8. Other Pre Specified Outcome: Number of Participants Reporting Complications Since Surgery
Description: Complications were collected by telephone interview after surgery.
Time Frame: Post-operative Day 1 Through 3 - Month Follow-up
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 54 | 51
Participants
  Operative extremity neurologic changes | 1 | 1 | 2
  Wound infection | 0 | 1 | 1
  Fall requiring medical attention | 1 | 2 | 1
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Operative extremity neurologic changes; Test type: Superiority; p = 0.843, Fisher Exact
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Wound infection; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 3: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Fall requiring medical attention; Test type: Superiority; p = 1.00, Fisher Exact

9. Other Pre Specified Outcome: Number of Participants Reporting a NRS Pain Score Greater Than 3
Description: as for outcome 1
Time Frame: 3 month follow up
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
Number analyzed (Participants) | 50 | 54 | 51
Participants
  Pain at rest | 0 | 1 | 1
  Pain with movement | 0 | 4 | 2
Statistical Analysis 1: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Pain at rest; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: PNB Bupivacaine vs PAI Ropivacaine vs PAI Liposomal Bupivacaine; Pain with movement; Test type: Superiority; p = 0.167, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of the study, from baseline through three month follow-up for each study participant.
Description: The Anesthesia Clinical Research Unit (ACRU) not affiliated with the investigator team had continuous access to information regarding adverse outcomes and monitored quarterly reporting to the principal investigator. Participants were postoperatively monitored for adverse outcomes by the inpatient pain service (IPS) or surgical team.
Arm/Group | PNB Bupivacaine | PAI Ropivacaine | PAI Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/51 | 3/54 | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNB Bupivacaine (N=51) | PAI Ropivacaine (N=54) | PAI Liposomal Bupivacaine (N=54)
Fall (General disorders) | 0 (0) | 0 (0) | 0 (0)
Nerve Injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Infection (General disorders) | 0 (0) | 0 (0) | 0 (0)
ICU admission (General disorders) | 0 (0) | 3 (3) | 0 (0)
Rapid response team (General disorders) | 0 (0) | 2 (2) | 0 (0)
Additional surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
PNB and PAI for total hip arthroplasty are highly technique dependent modalities and standardized delivery of PAI injections is less established than PNB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes